CLINICAL TRIAL: NCT04438226
Title: Surgical Approach of Hemiarthroplasty After Femoral Neck Fracture: Posterolateral or Direct Lateral
Acronym: APOLLO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: JointResearch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL63378.100.17
Record Dates: First submitted 2019-06-11; First posted 2020-06-18 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Hip Fractures; Surgical Approach; Hemiarthroplasty; Posterolateral; Direct Lateral
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Posterolateral (Experimental): Patients treated with a hemiarthroplasty using the posterolateral approach
  Interventions: Procedure: Surgical approach
- Direct lateral (Experimental): Patients treated with a hemiarthroplasty using the direct lateral approach
  Interventions: Procedure: Surgical approach

INTERVENTIONS:
Procedure: Surgical approach — The surgical approach of hemiarthroplasty after femoral neck fracture

SUMMARY:
Rationale: In the Netherlands the two main surgical approaches for hemiarthroplasty are the posterolateral and the direct lateral approach. Currently there is no conclusive evidence which of these two approaches results in better patient outcomes.

Objective: Assessing the patient outcome comparing the posterolateral with the direct lateral approach in patients being treated with cemented hemiarthroplasty after femoral neck fractures.

Study design: A randomised controlled multi-center superiority trial and natural experiment with an economic evaluation alongside.

Study population: All patients older than 18 years with a femoral neck fracture whereby treatment with cemented hemiarthroplasty is recommended according the national guidelines.

Intervention: Treatment with cemented hemiarthroplasty using the posterolateral approach.

Standard intervention to be compared to: Treatment with cemented hemiarthroplasty using the direct lateral approach.

Main study parameters/endpoints: The primary outcome is the patient-rated quality of life (EQ-5D-5L) at 6 months after surgery.

Secondary outcomes are: ADL functionality (KATZ), Balance test (SPPB), Tendency to Fall (FES-I), Pain (NRS), Re-interventions, Mobility, Discharge destination, Complications, and cost-effectiveness.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The different approaches in the two treatment arms of the randomised controlled trial are widely used techniques in the Netherlands and many of the outcome measures are part of the standard clinical follow-up after hip fracture. Therefore, there is no extra risk or burden for participating patients, except for the time to complete some additional follow-up measurements. The primary outcome measurement and secondary outcomes, will be assessed through questionnaires online, by hardcopy or by phone at baseline, 4 weeks, 3 and 6 months postoperatively. The assessment of the Short Physical Performance Battery (SPPB) balance test, will be performed by one of the study researchers or nurse practitioner to protect continuity and feasibility.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years at time of trauma
* Acute hip fracture
* Hemiarthroplasty as recommended treatment according the national guidelines
* Dutch or English fluency and literacy
* Informed consent or by proxy in patients with mental impairment

Exclusion Criteria:

* Multi-trauma-patient (ISS > 15)
* Secondary surgery after failed internal fixation
* Patients with a known metastatic disease and a confirmed pathological fracture of the hip
* Fracture > 7 days at time of surgery
* High risk of non-compliance/adherence to study procedures (e.g. no Dutch residency during follow-up period, or other factors that impair follow-up data collection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 555 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
EQ-5D-5L | at 6 months after surgery
  The EQ-5D-5L descriptive system assesses health in five dimensions (MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN / DISCOMFORT, ANXIETY / DEPRESSION), each of which has five levels of response (no problems, slight problems, moderate problems, severe problems, extreme problems/unable to). This part of the EQ-5D questionnaire provides a descriptive profile that can be used to generate a health state profile. Health state index scores generally range from less than 0 (where 0 is the value of a health state equivalent to dead; negative values representing values as worse than dead) to 1 (the value of full health), with higher scores indicating higher health utility. The second part of the questionnaire consists of a visual analogue scale (VAS) on which the patient rates his/her perceived health from 0 (the worst imaginable health) to 100 (the best imaginable health).

SECONDARY OUTCOMES:
Re-interventions | at 6 months after surgery
  Number of patients which are undergoing a re-intervention in the first 6 months after surgery
SPPB | at 4 months after surgery
  Balance test (SPPB)
FES-I | at 6 months after surgery
  The Falls Efficacy Scale-International (FES-I) is a short, easy to administer tool that measures the level of concern about fallingduring 16 social and physical activities inside and outside the home whether or not the person actually does the activity. The minimum score is 16 (no concern about falling) to the maximum score of 64 (severe concern about falling).
NRS | at 6 months after surgery
  Numeric Rating Scale (NRS) is a numeric scale to assess pain. The minimum score is 0 (no pain) and the maximum score is 10 (the worst imaginable pain)
KATZ | at 6 months after surgery
  Katz Index of Independence in Activities of Daily Living (ADL) is an instrument to assess functional status as a measurement of the client's ability to perform activities of daily living independently. The Index ranks adequacy of performance in the six functions of bathing, dressing, toileting, transferring, continence, and feeding. Clients are scored yes/no for independence in each of the six functions. A score of 6 indicates full function, 4 indicates moderate impairment, and 2 or less indicates severe functional impairment.
Mobility | at 6 months after surgery
  Mobility according to the mobility score. We'll assess the mobility according to the following options: no walking aids, 1 walking stick, walker or two crutches, in-house mobility but outside no mobility without aids, no functional mobility
Complications | During admission, 3 and 6 months post-operative
  The number of post-operative complications
Discharge destination | After admission, at 3 and 6 months post-operative
  Discharge destination: We'll ask where the patient is going to live after discharge, which we compare with the place where the patient was living before the trauma. The options are: independently at home, at home with care, nursing home, rehabilitation center.
Cost-effectiveness | at 4 weeks, 3 and 6 months post-operative
  An economic evaluation will be performed for physical functioning and Quality Adjusted Life Years (QALYs). For estimating QALYs, the patients' EQ-5D-5L health states will be converted into utility scores using the Dutch tariff. QALYs will subsequently be calculated using linear interpolation between measurement points.

CONTACTS AND LOCATIONS:
Locations (1):
- Onze Lieve Vrouwe Gasthuis, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tol MCJM, Willigenburg NW, Rasker AJ, Willems HC, Gosens T, Heetveld MJ, Schotanus MGM, Eggen B, Kormos M, van der Pas SL, van der Vaart AW, Goslings JC, Poolman RW; APOLLO Research Group. Posterolateral or Direct Lateral Surgical Approach for Hemiarthroplasty After a Hip Fracture: A Randomized Clinical Trial Alongside a Natural Experiment. JAMA Netw Open. 2024 Jan 2;7(1):e2350765. doi: 10.1001/jamanetworkopen.2023.50765. PMID 38206628